CLINICAL TRIAL: NCT03322553
Title: Endoscopic Full Thickness Plication (GERD-X) for the Treatment of PPI Dependent GERD: Randomized, Double Blinded, Sham Controlled Trial
Brief Title: Endoscopic Full Thickness Plication (GERD-X) for the Treatment of PPI Dependent GERD:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh K, Principal Investigator, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GERDX01
Record Dates: First submitted 2017-10-17; First posted 2017-10-26 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-10

CONDITIONS: Gastro Esophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomized, Double blinded, sham controlled trial
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plication group (Experimental): In patients allocated to endoscopic plication, endoscopic full-thickness plication will be performed using the GERDX® system. All procedures will be performed under general anesthesia. Savary-guidewire will be placed into the stomach using a gastroscope. The GERDX® system will be introduced over the guidewire into the stomach and retroflexed. The GE junction will be visualized using another slim endoscope passed through a channel present in the GERD-X device. According to study protocol, at least 2 pretied transmural pledgeted sutures will be deployed to achieve a tight closure of GE junction around the GERD-X device
  Interventions: Device: GERD-X
- Sham Group (Sham Comparator): In sham procedure, identical technique will be followed by positioning the plicator inside the stomach but sutures will not be applied.
  Interventions: Device: GERD-X

INTERVENTIONS:
Device: GERD-X — Endoscopic full-thickness plication will be performed using the GERDX® system. All procedures will be performed under general anesthesia. Savary-guidewire will be placed into the stomach using a gastroscope. The GERDX® system will be introduced over the guidewire into the stomach and retroflexed. The GE junction will be visualized using another slim endoscope passed through a channel present in the GERD-X device. According to study protocol, at least 2 pretied transmural pledgeted sutures will be deployed to achieve a tight closure of gastro-esophageal junction around the GERD-X device.

SUMMARY:
Gastro-esophageal reflux disease (GERD) is a common gastrointestinal disorder with a significant proportion of patients becoming dependent on proton pump inhibitor (PPI) therapy. Long term use of PPI therapy can be associated with side effects such as osteoporosis, small intestinal bacterial overgrowth and renal failure. Moreover, some of the patients might be reluctant to take PPIs for long duration and prefer surgery over pharmacotherapy. Endoscopic plication (GERD-X) is an alternative and less invasive procedure compared to laparoscopic fundoplication for the treatment of GERD. In endoscopic plication, transmural sutures are applied at the gastro-esophageal (GE) junction thereby reconstructing the gastric cardia and accentuating the valvular mechanism to prevent reflux. Only few trials have evaluated the efficacy of endoscopic plication technique and reported encouraging results. In this study we aim to evaluate the efficacy of a similar endoscopic technique but with application of two transmural sutures in randomized controlled method.

DETAILED DESCRIPTION:
Patients screening and inclusion:

The study will be conducted over 6-month period. Data of patients presenting with PPI dependent GERD will be recorded and maintained. At initial screening, GERD health related quality of life questionnaire (GERD HRQL) and requirement of anti-secretory medicines (detailed drug history) will be assessed along with gastroscopy. All anti-secretory medicines will be stopped for 7 days and GERD HRQL will be reassessed off drugs. Esophageal high resolution manometry with 24-h pH impedance monitoring will be done on the 8th day after stopping medicines. Basal lower esophageal sphincter (LES) pressure, esophageal motility pattern, 24-h esophageal acid exposure, non acidic bolus reflux, number of reflux episodes, DeMeester score, symptom index and symptom association probability would be assessed. Those patients with pathologic esophageal acid exposure (esophageal pH <4 for >4.2% of 24-h period) will be included in the trial. Patients will then be randomly assigned by a computer to either GERD-X or sham procedure with a target ratio of 1:1. The patient, principle investigator and the study coordinators would be blinded to the treatment assignment.

Intervention:

In patients allocated to endoscopic plication, endoscopic full-thickness plication will be performed using the GERDX® system. All procedures will be performed under general anesthesia. Savary-guidewire will be placed into the stomach using a gastroscope. The GERDX® system will be introduced over the guidewire and into the stomach. The subsequent procedure will be performed as described in previous studies, using a similar device (NDO Plicator). According to study protocol, at least 2 pretied transmural pledgeted sutures will be deployed to achieve a tight closure of GE junction around the endoscope. In sham procedure, identical technique will be followed by positioning the plicator 1cm below the GE junction but sutures will not be deployed.

Post intervention monitoring:

Immediately after the intervention, patients would be placed on soft diet and on demand analgesics for 5 days. Twice daily PPI will be given for all patients and would be stopped after 7 days. Thereafter, if patient experiences reflux symptoms, sucralfate, H2 blocker and PPI would be started sequentially in case of no response to the former drug after a period of 7days of therapy on each drug. Requirement and reintroduction of drugs will be enquired over phone and recorded appropriately.

Follow up:

Follow up visits will be carried out at 3, 6 and 12 months. During each visit, gastroscopy will be done to assess the gastro-esophageal junction along with evaluation of GERD HRQL and requirement of PPI. At 3 months post intervention, esophageal manometry and 24-h pH impedance monitoring would be performed.

Primary outcomes:

Improvement in GERD HRQL by more than 50% from baseline at 3 months

Secondary outcomes:

Improvement in GERD HRQL at 3, 6 and 12 months Improvement in symptom score and requirement of PPI at 3, 6 and 12 months Improvement in esophageal acid exposure and lower esophageal sphincter pressure at 3 months

Statistical Analysis The trial was designed to have a 90% power to detect a difference in GERD-HRQL post intervention at 5% level of significance.

The rate of improvement in GERD-HRQL for sham group is 35% and for active group is 70 %. A sample size of 38 is required for each group to achieve a statistical power of 80% at 5% type I error.

Statistical methods Continuous data will be expressed as median and inter-quartile range (IQR). Frequency will be expressed as percentage (%). Continuous and categorical data between active and sham groups will be compared using Mann-Whitney U test and Chi-square test, with Yates' correction as applicable, respectively. P values below 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients (between 18 to 60 years of age) with PPI dependent GERD and pathologic esophageal acid exposure as documented by percentage time esophageal pH less than 4 of more than 4.2% on pH-metry during 24-h period while off PPI
* Patients who are willing to pay the expenses of the GERD-X procedure

Exclusion Criteria:

* Large Hiatal hernia >3cm
* Gr C/D esophagitis
* Lower esophageal sphincter (LES) pressure <5 or >15 mm Hg
* Paraesophageal hernia
* GE flap valve grade IV (Hill's classification)
* Barretts esophagus
* Esophageal dysmotility
* ASA physical status >II
* Previous esophageal or gastric surgery
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Improvement in GERD | 3months
  Improvement in GERD HRQL by more than 50% from baseline at 3 months
  GERD - Health Related Quality of Life Questionnaire (GERD-HRQL) :
  Total Score: Calculated by summing the individual scores toquestions 1-15 Greatest possible score ( worst symptoms)= 75 Lowest possible score ( no symptoms)= 0
  Heartburn Score: Calculated by summing the individual scores to questions 1-6 .
  Worst heartburn symptoms = 30 No heartburn symptoms= 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination.
  Regurgitation Score: Calculated by summing the individual scores to questions10-15.
  Worst regurgitation symptoms = 30 No regurgitation symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.

SECONDARY OUTCOMES:
Improvement in GERD overall symptom and quality of life score | 12 months
  Improvement in GERD HRQL at 3, 6 and 12 months
  GERD - Health Related Quality of Life Questionnaire (GERD-HRQL) :
  Total Score: Calculated by summing the individual scores toquestions 1-15 Greatest possible score ( worst symptoms)= 75 Lowest possible score ( no symptoms)= 0
  Heartburn Score: Calculated by summing the individual scores to questions 1-6 .
  Worst heartburn symptoms = 30 No heartburn symptoms= 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination.
  Regurgitation Score: Calculated by summing the individual scores to questions10-15.
  Worst regurgitation symptoms = 30 No regurgitation symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.
Improvement in GERD symptom sub-score | 12 months
  Improvement in GERD symptom (heartburn and regurgitation) score at 3, 6 and 12 months
  GERD - Health Related Quality of Life Questionnaire (GERD-HRQL) :
  Total Score: Calculated by summing the individual scores toquestions 1-15 Greatest possible score ( worst symptoms)= 75 Lowest possible score ( no symptoms)= 0
  Heartburn Score: Calculated by summing the individual scores to questions 1-6 .
  Worst heartburn symptoms = 30 No heartburn symptoms= 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination.
  Regurgitation Score: Calculated by summing the individual scores to questions10-15.
  Worst regurgitation symptoms = 30 No regurgitation symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.
Requirement of PPI | 12 months
  Requirement of PPI for control of symptoms at 3, 6 and 12 months
  Heartburn and Regurgitation questionnaire
  0 =No symptom
  1 =Symptoms noticeablebut not bothersome 2=S ymptoms noticeableand bothersome but noteve ry day 3 =Symptoms bothersome every day 4 =Symptoms affect daily activity 5 =Symptoms are incapacitating to do daily activities
Improvement in oesophageal acidification | 3 months
  Improvement in oesophageal acid exposure at 3 months
  pH more than 4 of more than 4.2%
Improvement in lower oesophageal sphincter pressure | 3 months
  Improvement in lower oesophageal sphincter pressure at 3 months
  Lower Esophageal Sphincter pressure > 15 mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Dr. D. Nageshwar Reddy, MBBS, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalapala R, Karyampudi A, Nabi Z, Darisetty S, Jagtap N, Ramchandani M, Gupta R, Lakhtakia S, Goud R, Venkat Rao G, Sharma P, Reddy DN. Endoscopic full-thickness plication for the treatment of PPI-dependent GERD: results from a randomised, sham controlled trial. Gut. 2022 Apr;71(4):686-694. doi: 10.1136/gutjnl-2020-321811. Epub 2021 Apr 13. PMID 33849942